CLINICAL TRIAL: NCT07139327
Title: A Pre-market, Prospective, Interventional, Multicenter, Pivotal Study to Evaluate Efficacy and Safety of a Totally Implantable Cochlear Implant System in an Adult Population With Sensorineural Hearing Loss
Brief Title: A Pivotal Study to Evaluate the Efficacy and Safety of a Totally Implantable Cochlear Implant (TICI) System in Adults
Acronym: ENTERPRISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5864
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hearing Loss, Bilateral Sensorineural
Keywords: cochlear implant; sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TICI G2 Clinical Investigation System (Experimental): Participants will be implanted with the TICI G2 Implant
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — TICI G2 Clinical Investigation System

SUMMARY:
This clinical study examines the performance of an investigational totally implantable cochlear implant (TICI) system. The system includes an implantable microphone under the skin to detect speech and sound from the environment allowing the option to hear without the need of an external sound processor. This implant will be tested in adults with sensorineural hearing loss, a type of hearing loss caused by damage to the inner ear or auditory nerve (the nerve that carries sound signals from the ear to the brain). The study participants will undergo a series of tests that include testing their implant and their hearing. They will also complete questionnaires to see how they rate their hearing and overall general health.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years and older at time of consent.
* Clinically established post-linguistic moderately severe to profound sensorineural hearing loss (PTA4 of >55 dB HL), in the ear to be implanted.
* Meets local candidacy criteria for cochlear implantation.
* Compromised functional hearing with a hearing aid in the ear to be implanted, as determined by the investigator.
* Willing to undergo unilateral cochlear implantation.
* Candidate is a fluent speaker in the language used to assess speech perception performance as determined by the investigator
* Direct access to a compatible Smart Phone.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Prior cochlear implantation, in either ear, or medical plan for cochlear implantation during the clinical investigation, contralateral to the ear to be implanted.
* Candidates with single-sided deafness as determined by the investigator.
* Intra-axial (within-the-brain) lesions or deafness due to lesions of the acoustic nerve affecting the ear to be implanted.
* Middle ear infection (including acute otitis media, chronic otitis media, suppurative otitis media, or serous drainage) in the ear to be implanted either at the time of surgery or within 3 months prior to enrolment.
* Presence of a tympanic membrane perforation or a history of otologic surgery within 3 months prior to enrolment, in the ear to be implanted.
* Previously reported diagnosis of auditory neuropathy, in the ear to be implanted.
* Cochlear ossification, cochlear malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, in the ear to be implanted.
* Current cerebrospinal fluid (CSF) shunts or drains, existing perilymph fistula, skull fracture or CSF leaks.
* Severe, or poorer, bilateral sensorineural hearing loss prior to 5 years of age, as reported by the participant.
* Severe, or poorer, sensorineural hearing loss for more than 20 years, as reported by the participant, in the ear to be implanted.
* Medical or psychological conditions that contraindicate general anaesthesia, surgery, or participation in the clinical investigation as determined by the investigator.
* Preexisting skin condition that could jeopardize wound healing, as determined by the investigator e.g., psoriasis, dermatitis, use of corticosteroids, uncontrolled diabetes.
* Unrealistic expectations on the part of the participant, regarding the possible benefits, risks, and limitations inherent to the surgical procedure(s) and prosthetic devices, as determined by the Investigator.
* Additional disabilities that may affect the subject's participation or safety during the clinical investigation.
* Women who are pregnant.
* Investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as spouse, parent, child or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of the investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator (unless Cochlear sponsored and determined by Investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Speech recognition performance in quiet | Preimplantation to 6 months post-activation
  Percent correct word score from preimplantation to post-activation
Incidence of adverse events and device deficiencies | Implantation to 6 and 12 months post-activation
  Frequency and severity of device and procedure-related adverse events, including device deficiencies

SECONDARY OUTCOMES:
Speech recognition in quiet and noise | Preimplantation to 12 months post-activation
  Percent correct scores for word tests in quiet and speech reception threshold scores for sentence tests in noise
Speech Spatial Qualities questionnaire (SSQ-12) | Preimplantation to 12 months post-activation
  Speech, Spatial, and Qualities of Hearing Scale Global score (SSQ-12). Scores range from 0 to 10, where higher scores indicate greater ability (less hearing disability).
Cochlear Implant Quality of Life Profile (CIQOL-35) | Preimplantation to 12-months post-activation
  Cochlear implant hearing related quality of life score (CIQOL-35). Scored for six health domains (communication, emotional, entertainment, environment, listening effort, and social) each scaled from 0 to 100, where a higher score indicates better health.
Health Utilities Index (HUI 2/3) | Preimplantation to 12 months post-activation
  Health Utilities Index (HUI 2/3) Global score. Scores range from -0.36 to 1.00, where a negative score represents a state "worse than dead" and a top score of 1.00 is "perfect health"
Living with Cochlear Implants Questionnaire (LivCI) | Preimplantation to 12 months post-activation
  Living with Cochlear Implants Questionnaire (LivCI) evaluates the impact of a hearing device on four domains, Participation (range 0 to 12), Psychosocial & Wellbeing (range 0 to 21), Stigma (range 0 to 15) and Management & Aesthetics (range 0 to 18), where a higher domain score indicates positive patient report.
Patient Satisfaction Survey | 6 to 12 months post-activation
  Device satisfaction rating score. Scores range from 1 to 5, where a higher score indicates greater patient satisfaction with the TICI system.
Short Form (SF)-36 Health Survey | 8 to 10 months post-activation
  SF-36 is scored for eight health domains, each scaled from 0 to 100, where a higher score indicates better health.
Time on air | Initial activation to 12 months post-activation
  Hours of TICI System usage

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Macquarie University Hospital, Macquarie, New South Wales
  - Westmead Private Hospital, Westmead, New South Wales
  - Westmead Public Hospital, Westmead, New South Wales
  - Royal Victoria Eye and Ear Hospital, East Melbourne, Victoria
  - St Vincent's Private Hospital, East Melbourne, Victoria
- France (2):
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Centre Hospitalier Universitaire de Lille, Lille

IPD SHARING:
Plan to Share IPD: No